CLINICAL TRIAL: NCT04141137
Title: TRICUS STUDY EURO - Safety and Efficacy of the TricValve® Transcatheter Bicaval Valves System in the Superior and Inferior Vena Cava in Patients With Severe Tricuspid Regurgitation
Brief Title: TRICUS STUDY Euro - Safety and Efficacy of the TricValve® Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: P+F Products + Features GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-TRIC-002
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Severe Tricuspid Regurgitation
Keywords: Tricuspid Valve Insufficiency; Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TricValve® System Single-Arm (Experimental): Two self-expanding biological valves for implantation into the inferior and superior vena cava.
  Interventions: Device: TricValve® System

INTERVENTIONS:
Device: TricValve® System — The TricValve® Delivery System (catheter) with already pre-mounted biological heart valve is inserted from the femoral vein to access the inferior vena cava (IVC) and superior vena cava (SVC) of the heart under fluoroscopy guidance. The appropriately sized TricValve® is released at the implantation site and positions itself as per the anatomy - self expanding frame.

SUMMARY:
The TricValve® Transcatheter Bicaval Valves System is indicated for relief of tricuspid insufficiency in patients with symptomatic heart disease who are judged by a heart team, including a cardiac surgeon, to be at extreme risk or inoperable for open surgical therapy.

DETAILED DESCRIPTION:
TricValve® Transcatheter Bicaval Valves is a system of two self-expanding biological valves for the treatment of patients with hemodynamically relevant tricuspid insufficiency and caval reflux. The prostheses are implanted percutaneously into the inferior and superior vena cava without disturbing the native tricuspid valve. It is especially intended for use for patients at extreme risk or who are inoperable for open surgical therapy. Pre-Clinical and Clinical preliminary studies have shown an acceptable safety and performance profile of the TricValve® Transcatheter Bicaval Valves System. Given that the medical device is a potential long-term treatment for patients with tricuspid insufficiency, clinical data for long-term treatment periods is necessary. Thus, the current study with the aim of CE certification is designed to investigate the safety and performance for at least 30 days and up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be 18 years of age or older
2. The subject must be a patient with severe symptomatic tricuspid regurgitation demonstrated by echocardiography with significant backflow in the lower (IVC) and/or upper (SVC) vena cava and with a v-wave ≥ 25 mmHg as demonstrated by right heart catheterization (measured in the IVC and/or SVC 2-4 cm above/ below RA inflow) within 8 weeks prior to the implantation
3. Suitable for TricValve® Transcatheter Bicaval Valves System implantation according to anatomic criteria by computed tomography
4. The subjects must have severe, tricuspid regurgitation leading to NYHA class III or IV
5. The subject has LVEF ≥ 40%
6. Distance covert in 6-minute walk test (6MWT) ≥ 60m
7. The patient shall be screened by a "Heart Team" - including an interventional cardiologist, cardiothoracic surgeon, and agreed as a candidate for TricValve® Transcatheter Bicaval Valves System implantation
8. Patient/authorized legal guardian understands the nature of the procedure, is willing to comply with associated follow-up evaluations, and provides written informed consent
9. Patient/patient's authorized legal guardian is geographically stable (or willing to return for required study follow-up) and understands and is willing to fulfil all of the expected requirements of this clinical protocol
10. Optimal medical treatment of patient

Exclusion Criteria:

1. Known significant intracardiac shunt (e.g. ventricular septal defect) or congenital structural heart disease based on heart teams decision
2. Requirement for other elective cardiac procedures e.g. PCI (percutaneous treatment of coronary artery) or CABG (coronary artery bypass surgery) up to 90 days after the procedure or 30 days before the procedure
3. Right ventricular failure (TAPSE ≤13mmHg)
4. Systolic pulmonary arterial pressure > 65 mmHg as assessed by Doppler echocardiography
5. Presence of any known life threatening (non-cardiac major or progressive disease), non-cardiac disease that will limit the subject's life expectancy to less than one year
6. Cerebro-vascular event within the past 3 months
7. History of mitral/tricuspid endocarditis within the last 12 months
8. Patient has untreated significant left sided valvular heart disease which requires treatment (e.g. mitral regurgitation or stenosis, and aortic regurgitation or stenosis)
9. Documented primary coagulopathy or platelet disorder, including thrombocytopenia (absolute platelet count <90k)
10. Documented evidence of significant renal dysfunction (serum creatinine > 3.0mg/dl) or on any form of dialysis at time of screening within the last 4 weeks
11. Contraindication or known allergy to device's components, anti-coagulation therapy with vitamin K antagonists or contrast media that cannot be adequately premedicated
12. Patients unsuitable for implantation because of thrombosis of the lower venous system or vena cava filter
13. The patient has contraindication against a transesophageal echo (TEE) during the procedure
14. Evidence of an acute myocardial infarction (AMI) ≤ 1 month (30 days)
15. Liver cirrhosis Child C (see appendix)
16. Female patient of child-bearing potential
17. Psychiatric or behavioural disease including known alcohol or drug abuser that is likely to impair compliance with protocol
18. Currently participating in another study of an investigational drug or device that would directly impact the treatment or outcome of the current study
19. Requirement for antibiotic treatment within the last 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with major adverse events | 30 days
  The percentage of participants with major adverse events (death, myocardial infarction, cardiac tamponade, cardiac surgery for failed TricValve® implantation, stroke. Major bleeding according to Valve Academic Research Consortium (VARC) criteria)
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 3 months
  Number of Patients with improvement in quality of life as assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ, a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Range of 0-100, in which higher scores reflect better health status.)

SECONDARY OUTCOMES:
Percentage of participants with major adverse events | up to 6 months
  The percentage of participants with major adverse events
Successful implantation | Up to Discharge (≤ 10 days post index procedure)
  The percentage of surviving participants with successful access, delivery and retrieval of the device delivery system, and deployment and correct positioning of the intended device(s), and no need for additional unplanned or emergency surgery or re-intervention related to the device or access procedure.
Unrestricted movement of cusps | Up to 30 days, up to 6 months
  The percentage of medical devices with unrestricted movement of cusps after implantation as assessed with echocardiography (nominal)
Cusp insufficiency | Up to 30 days, up to 6 months
  The change of the degree of cusp insufficiency as assessed with echocardiography (ordinal) from a higher to a lower value
Device success | Up to 30 days, up to 6 months
  Device success as measured by number of patients who are alive with intended device in place with no additional surgical or interventional procedures related to the TricValve®.
NYHA functional class | Up to 30 days
  Change of New York Heart Association (NYHA) functional class from III or IV to a lower one
6 Minute Walk Test | Up to 30 days, up to 6 months
  Improvement in distance (m) in the 6 Minute Walk Test
Kansas City Cardiomyopathy Questionnaire (KCCQ) | Up to 6 months
  Number of Patients with improvement in quality of life as assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ, a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Range of 0-100, in which higher scores reflect better health status.)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lauten, Prof.Dr.med., Principal Investigator — Charite University, Berlin, Germany; Iniguez Romo Andrés, Dr., Principal Investigator — Hospital Universitario Alvaro Cunqueiro- Vigo; Christian Hengstenberg, UnivProf.Dr., Principal Investigator — Medical University of Vienna
Locations (10):
- Austria (2):
  - Medizinische Universität Wien, Vienna
  - Krankenhaus Nord - Klinik Floridsdorf, Vienna
- Spain (8):
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Universitario Reina Sofia de Córdoba, Córdoba
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Universitario Alvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: No